CLINICAL TRIAL: NCT00679497
Title: A Phase I Study of MVA-B in Healthy Volunteers at Low Risk of HIV Infection
Brief Title: A Phase I Study of Modified Vaccinia Virus Ankara (MVA-B) in Healthy Volunteers at Low Risk of HIV Infection
Acronym: RisVac02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RisVac02; EudraCT: 2007-002367-27
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: Low risk HIV infection; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): MVA HIV-B
  Interventions: Biological: MVA-B
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MVA-B — * Modified Pox virus, strain MVA clade -B (expressing HIV-1 Bx08gp120 and IIIB gagpolnef)
    -~ 1 x 10e8 pfu/ml
  * 3 immunisations at week 0, 4 and 16
  Arms: 1
Biological: Placebo — -3 immunisations at week 0, 4 and 16
  Arms: 2

SUMMARY:
The purpose of this clinical trial is to study a modified pox viral vector considering:

1. HIV subtype B accounts for the most frequent virus strain in Europe and North America, as well as in many parts of the world.
2. This novel vaccinia construct expressing HIV subtype B gag, pol, env and nef antigens is to be studied in humans for the first time.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age between 18 and 55 years on the day of screening
* available for follow-up for the duration of the study (52 weeks from screening)
* able to give written informed consent
* at low risk of HIV and willing to remain so for the duration of the study low risk of HIV infection defined as: no history of injecting drug use in the previous ten years no gonorrhoea or syphilis in the last six months no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months no unprotected anal intercourse in the last six months no unprotected vaginal intercourse outside a relationship with a regular known/presumed HIV negative partner in the last six months
* willing to undergo a HIV test
* willing to undergo a genital infection screen
* if heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable contraceptive; IUCD; consistent record with condoms if using these; physiological or anatomical sterility in self or partner) from 14 days prior to the first vaccination until 4 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination
* if heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination

Exclusion Criteria:

* positive for hepatitis B surface antigen, hepatitis C antibody, antibody responses to vaccinia or serology indicating active syphilis requiring treatment
* pregnant or lactating
* clinically relevant abnormality on history or examination including history of grand-mal epilepsy, severe eczema, immunodeficiency or use of immunosuppressives in preceding 3 months
* receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of enrolment
* receipt of blood products or immunoglobin within 4 months of screening
* participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
* history of severe local or general reaction to vaccination defined as local: extensive, indurated redness and swelling involving most of the front-lateral thigh or the major circumference of the arm, not resolving within 72 hours general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal
* HIV 1/2 positive or indeterminate on screening
* positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
* grade 1 routine laboratory parameters
* unlikely to comply with protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety: proportion of patients with Grade 3 or above local, systemic or other clinical or laboratory adverse events. Adverse events attributable to discontinuation of the immunisation regimen. Immunogenicity: cellular responses (ELISPOT) | Safety: at any point of the study; Immunogenicity:week 6/8, 18/20, and at any point following immunisations

SECONDARY OUTCOMES:
Proportion of patients with grade 1 and 2 adverse events within 28 days of a vaccination -antibody responses -cellular responses -intracellular cytokine analysis | at any point of the study and at week 6 and 18 for intracellular cytokine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Gatell, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid

REFERENCES:
- [Result] Garcia F, Bernaldo de Quiros JC, Gomez CE, Perdiguero B, Najera JL, Jimenez V, Garcia-Arriaza J, Guardo AC, Perez I, Diaz-Brito V, Conde MS, Gonzalez N, Alvarez A, Alcami J, Jimenez JL, Pich J, Arnaiz JA, Maleno MJ, Leon A, Munoz-Fernandez MA, Liljestrom P, Weber J, Pantaleo G, Gatell JM, Plana M, Esteban M. Safety and immunogenicity of a modified pox vector-based HIV/AIDS vaccine candidate expressing Env, Gag, Pol and Nef proteins of HIV-1 subtype B (MVA-B) in healthy HIV-1-uninfected volunteers: A phase I clinical trial (RISVAC02). Vaccine. 2011 Oct 26;29(46):8309-16. doi: 10.1016/j.vaccine.2011.08.098. Epub 2011 Sep 9. PMID 21907749